CLINICAL TRIAL: NCT02660463
Title: Prospective Registry to Evaluate the Effective Incidence of Chronic Thromboembolic Pulmonary Hypertension in Germany
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kerckhoff Klinik (Other)
Collaborators: Hannover Medical School (Other); University Hospital, Saarland (Other)
Responsible Party: Principal Investigator, Dr. Thorsten Kramm, Dr. Thorsten Kramm, M.D., Kerckhoff Klinik
Other Study IDs: CTEPH-2016
Record Dates: First submitted 2016-01-12; First posted 2016-01-21 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: CTEPH; Chronic Thromboembolic Pulmonary Hypertension
Keywords: incidence; risk factors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Registration of the diagnosis "CTEPH" — Registration of risk factors for thromboembolic events

SUMMARY:
The incidence of chronic thromboembolic pulmonary hypertension (CTEPH) after acute pulmonary embolism ist not clear. It is estimated to be up to 3.8%. Prospective data registration does not exist. Treatment of choice is pulmonary endarterectomy if the thromboembolic lesions are surgically accessible. Otherwise interventional therapy by means of pulmonary balloon-angioplasty (BPA) or medical therapy is indicated. In Germany, the majority of the patients is referred to three CTEPH centers: Kerckhoff Clinic, Saarland University Hospital and Hannover Medical School to evaluate the therapeutic options. Starting in January 2016 all incident patients will be de-identified and included prospectively. Risk factors, outcome and treatment will be documented.

DETAILED DESCRIPTION:
All patients referred to the participating centers will be diagnosed in a standardized manner to confirm the diagnosis "CTEPH". No additional intervention or blood sampling is necessary. The recommended treatment option is the result of weekly CTEPH conferences. Every patient will be discussed.

The registry contains the following data:

Center PLZ Sex Age Body Mass Index History of venous thromboembolism (VTE), Date ff 1st VTE Anticoagulation and type of anticoagulation Blood group V/Q scan CT-agiography Pulmonary angiogram World Health Organisation-Functional Class six-minute walk distance Right heart catheter: RAP, PAPs, PAPd, PAPm, PAWP, CO, CI, PVR, SvO2 Treatment: PEA, Ballon Pulmonary Angioplasty (BPA), medically therapy, Vena cava filter CTEPH special risk factors: thrombophilia, antiphospholipid antibody syndrome, splenectomy, VA shunt; pacemakers

ELIGIBILITY:
Inclusion Criteria:

* diagnosis "CTEPH" confirmed

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient with confirmed CTEPH during the year 2016 or not diagnosis confirmation not more than 6 months ago
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Diagnosis "CTEPH" confirmed | 12 months
  Aim of the study is to detect prospectively the incidence of the diagnosis CTEPH during one year in Germany.
Treatment | 12 months
  Registration of the frequency of different treatment options, e.g. pulmonary endarterectomy, pulmonary ballon-angioplasty and medical therapy

CONTACTS AND LOCATIONS:
Overall Officials: Eckhard Mayer, Prof. Dr., Study Chair — Kerckhoff Klinik, Bad Nauheim, Germany
Locations (2):
- Germany (2):
  - Kerckhoff Clicic, Bad Nauheim
  - Hannover Medical School, Hanover

REFERENCES:
- [Background] Condliffe R, Kiely DG, Gibbs JS, Corris PA, Peacock AJ, Jenkins DP, Goldsmith K, Coghlan JG, Pepke-Zaba J. Prognostic and aetiological factors in chronic thromboembolic pulmonary hypertension. Eur Respir J. 2009 Feb;33(2):332-8. doi: 10.1183/09031936.00092008. Epub 2008 Oct 1. PMID 18829679
- [Background] Condliffe R, Kiely DG, Gibbs JS, Corris PA, Peacock AJ, Jenkins DP, Hodgkins D, Goldsmith K, Hughes RJ, Sheares K, Tsui SS, Armstrong IJ, Torpy C, Crackett R, Carlin CM, Das C, Coghlan JG, Pepke-Zaba J. Improved outcomes in medically and surgically treated chronic thromboembolic pulmonary hypertension. Am J Respir Crit Care Med. 2008 May 15;177(10):1122-7. doi: 10.1164/rccm.200712-1841OC. Epub 2008 Feb 21. PMID 18292468
- [Background] McGoon MD, Benza RL, Escribano-Subias P, Jiang X, Miller DP, Peacock AJ, Pepke-Zaba J, Pulido T, Rich S, Rosenkranz S, Suissa S, Humbert M. Pulmonary arterial hypertension: epidemiology and registries. J Am Coll Cardiol. 2013 Dec 24;62(25 Suppl):D51-9. doi: 10.1016/j.jacc.2013.10.023. PMID 24355642
- [Result] Wilkens H, Lang I, Behr J, Berghaus T, Grohe C, Guth S, Hoeper MM, Kramm T, Kruger U, Langer F, Rosenkranz S, Schafers HJ, Schmidt M, Seyfarth HJ, Wahlers T, Worth H, Mayer E. Chronic thromboembolic pulmonary hypertension (CTEPH): updated Recommendations of the Cologne Consensus Conference 2011. Int J Cardiol. 2011 Dec;154 Suppl 1:S54-60. doi: 10.1016/S0167-5273(11)70493-4. PMID 22221974
- [Derived] Kramm T, Wilkens H, Fuge J, Schafers HJ, Guth S, Wiedenroth CB, Weingard B, Huscher D, Pittrow D, Cebotari S, Hoeper MM, Mayer E, Olsson KM. Incidence and characteristics of chronic thromboembolic pulmonary hypertension in Germany. Clin Res Cardiol. 2018 Jul;107(7):548-553. doi: 10.1007/s00392-018-1215-5. Epub 2018 Feb 15. PMID 29450722